CLINICAL TRIAL: NCT04336982
Title: An Exploratory Phase 1b Open-label Multi-arm Trial to Evaluate the Safety and Efficacy of CC-90009 in Combination With Anti-Leukemia Agents in Subjects With Acute Myeloid Leukemia
Brief Title: A Safety and Efficacy Study of CC-90009 Combinations in Subjects With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90009-AML-002; U1111-1247-5619 (Other: WHO); 2019-001681-15 (EudraCT Number)
Record Dates: First submitted 2020-03-26; First posted 2020-04-07 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: CC-90009; Venetoclax; Azacitidine; Gilteritinib; Hematologic cancers; Leukemia; Acute myeloid leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — CC-90009; venetoclax; Azacitidine; gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CC-90009 in combination with venetoclax and azacitidine (Experimental): CC-90009 will be administered intravenously per dosing schedule in a 28-day cycle. Venetoclax will be administered orally QD.
  Azacitidine will be administered intravenously or subcutaneously on planned dosing days for each cycle.
  Interventions: Drug: CC-90009; Drug: Venetoclax; Drug: Azacitidine
- CC-90009 in combination with gilteritinib (Experimental): CC-90009 will be administered intravenously per dosing schedule in a 28-day cycle. Gilteritinib will be administered orally QD.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: CC-90009 — Injection
  Arms: CC-90009 in combination with venetoclax and azacitidine
Drug: Venetoclax — Tablet
  Arms: CC-90009 in combination with venetoclax and azacitidine
Drug: Azacitidine — Injection
  Arms: CC-90009 in combination with venetoclax and azacitidine
Drug: Gilteritinib — Tablet
  Arms: CC-90009 in combination with gilteritinib

SUMMARY:
CC-90009-AML-002 is an exploratory Phase 1b, open-label, multi-arm trial to evaluate the safety and efficacy of CC-90009 in combination with anti-leukemia agents in participants with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Study CC-90009-AML-002 is an open-label, multi-arm, parallel multi-cohort, multicenter, Phase 1b study to determine the safety, tolerability, PK, and efficacy of CC 90009 in combination with anti-leukemia agents used for the treatment of AML. CC 90009 will be given as a combination therapy to subjects with newly diagnosed (ND) or relapsed or refractory (R/R) AML.

The dose and schedule finding part (Part A) of the study will evaluate the safety, PK and PD data, and preliminary efficacy information and determine the Part B dose and schedule for each arm.

The expansion part (Part B) of the study will further evaluate the safety and efficacy of the CC-90009 containing combination at or below the maximum tolerated dose (MTD) in the selected cohorts in order to determine the recommended Phase 2 dose (RP2D) for subjects with AML.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
2. Arm A (CC-90009 + venetoclax/azacitidine):

   1. Part A: Newly diagnosed AML with poor/adverse risk genetic abnormalities and is either ≥ 75 years of age or is ineligible for intensive chemotherapy OR
   2. Part A: Primary Refractory AML, or AML in first relapse, and is ≥ 18 years of age
   3. Part B: Newly diagnosed AML and is ≥ 75 years of age or intensive chemotherapy ineligible
3. Arm B (CC-90009 + gilteritinib):

   1. Subject is ≥ 18 years of age.
   2. Fms-like tyrosine kinase 3 (FLT3) mutation positive.
   3. Gilteritinib treatment naïve
4. Subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Subject must have the following screening laboratory values:

   * Total White Blood Cell count (WBC) < 25 x 10^9/L prior to study treatments. Treatment with hydroxyurea to achieve this level is allowed.
   * Selected electrolytes within normal limits or correctable with supplements.

     * Participant must have adequate liver function as demonstrated by: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) and bilirubin ≤ 1.5 x ULN
     * Participant has adequate renal function as demonstrated by an estimated serum creatinine clearance of ≥ 30 mL/min.
6. Agree to follow the CC-90009 Pregnancy Prevention Plan (PPP) and combination agents' requirements.

Exclusion Criteria:

1. Subject with acute promyelocytic leukemia (APL)
2. Subject has received systemic anticancer therapy (including investigational therapy) or radiotherapy < 28 days or 5 half-lives, whichever is shorter, prior to the start of study treatment
3. Patients with prior autologous hematopoietic stem cell transplant (HSCT) who, in the investigator's judgment, have not fully recovered from the effects of the last transplant (eg, transplant related side effects)
4. Prior allogeneic HSCT with either standard or reduced intensity conditioning ≤ 6 months prior to dosing
5. Subject on systemic immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). The use of topical steroids for ongoing skin or ocular GVHD is permitted
6. Subject has persistent, clinically significant non-hematologic toxicities from prior therapies which have not recovered to < Grade 2
7. Subject has or is suspected of having central nervous system (CNS) leukemia. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening.
8. Disorders or conditions disrupting normal calcium homeostasis or preventing calcium supplementation.
9. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. Left ventricular ejection fraction (LVEF) < 45% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO).
   2. Complete left bundle branch or bifascicular block.
   3. Congenital long QT syndrome.
   4. Persistent or clinically meaningful ventricular arrhythmias.
   5. QTcF ≥ 470 ms (Arm A) or > 450 ms (Arm B) on Screening electrocardiogram (ECG)
   6. Unstable angina pectoris or myocardial infarction ≤ 6 months prior to starting study treatments or unstable arrhythmia.
   7. Cardiovascular disability status of New York Heart Association Class ≥2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
10. Subject is a pregnant or lactating female
11. Additional exclusion criteria based on combination agent:

    a. For Combination Arm A (venetoclax/azacitidine):
    * Received strong or moderate CYP3A inhibitors or inducers or P-gp inhibitors within 7 days prior to initiation of first venetoclax dose.
    * Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or Star fruit within 3 days prior to first venetoclax dose through last dose of venetoclax.
12. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to C1D1.

    a. Acute symptoms must have resolved and based on investigator assessment in consultation with the medical monitor, there are no sequelae that would place the participant at a higher risk of receiving study treatment.
13. Previous SARS-CoV-2 vaccine within 14 days of C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 28 days
  Number of participants with a DLT
Adverse Events (AEs) | Up to 28 days after last dose of study drug.
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology.

SECONDARY OUTCOMES:
Complete Remission Rate (CRR), | Up to 3 years
  is defined as the rate for any type of CR or CRh
Objective Response Rate (ORR) | Up to 3 years
  includes all responses of complete remissions (CRs), Morphologic leukemia-free state (MLFS), and Partial remission (PR)
Progression Free Survival (PFS) | Up to 3 years
  is defined as the time from the first dose of study drug(s) to the first occurrence of relapse or progression or death from any cause
Overall Survival (OS) | Up to 3 years
  is measured as the time from the first dose of study drug(s) to death due to any cause and will be analyzed in a manner similar to that described for PFS.
Duration of Remission | Up to 3 years
  is measured from the time when criteria for CR/CRh/PR are first met (whichever is first recorded) until the first date at which relapse, or progressive disease is objectively documented.
Time to Remission | Up to 3 years
  is measured from the time when criteria for CR/CRh/PR are first met (whichever is first recorded)
Pharmacokinetics - Cmax | Until last CC-90009 dose in Cycle 3 (each cycle is 28 days. CC-90009 dosing days are Days 1-5 in Cycle 3)
  observed maximum concentration in plasma
Pharmacokinetics - AUC24 | Until last CC-90009 dose in Cycle 3 (each cycle is 28 days. CC-90009 dosing days are Days 1-5 in Cycle 3)
  area under the plasma concentration time-curve from time 0 to 24 hours postdose
Pharmacokinetics - t1/2 | Until last CC-90009 dose in Cycle 3 (each cycle is 28 days. CC-90009 dosing days are Days 1-5 in Cycle 3)
  terminal half life

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (7):
  - Local Institution - 104, San Francisco, California
  - Local Institution - 107, New Haven, Connecticut
  - Local Institution - 103, Boston, Massachusetts
  - Local Institution - 101, St Louis, Missouri
  - Local Institution - 108, Hackensack, New Jersey
  - Local Institution - 105, Houston, Texas
  - Local Institution - 102, Seattle, Washington
- Local Institution - UNK3, Yvoir, Belgium
- Canada (2):
  - Local Institution - 202, Edmonton, Alberta
  - Local Institution - 201, Toronto, Ontario
- France (3):
  - Local Institution - 402, Marseille
  - Local Institution - 401, Pessac
  - Local Institution - 404, Toulouse
- Local Institution - 301, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Surka C, Jin L, Mbong N, Lu CC, Jang IS, Rychak E, Mendy D, Clayton T, Tindall E, Hsu C, Fontanillo C, Tran E, Contreras A, Ng SWK, Matyskiela M, Wang K, Chamberlain P, Cathers B, Carmichael J, Hansen J, Wang JCY, Minden MD, Fan J, Pierce DW, Pourdehnad M, Rolfe M, Lopez-Girona A, Dick JE, Lu G. CC-90009, a novel cereblon E3 ligase modulator, targets acute myeloid leukemia blasts and leukemia stem cells. Blood. 2021 Feb 4;137(5):661-677. doi: 10.1182/blood.2020008676. PMID 33197925
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html